CLINICAL TRIAL: NCT06727695
Title: A Comparative Study of Training Effectiveness: Technogyms Biostrength Devices Vs. Conventional Strength Training Devices: a Randomized Controlled Trial
Brief Title: Effect of BioStrength Training on Muscle Strength and Satisfaction in Adults Aged 30-65
Acronym: BIO-STR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio-RCT-2024-01
Record Dates: First submitted 2024-09-30; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Muscle Strength; Body Composition; Physical Fitness
Keywords: Strength training; Muscle strength; Body composition; Customer satisfaction; BioStrength; Technogym; Resistance training; Fitness equipment; Handgrip strength; Randomized controlled trial
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No BioStrength Training) (Active Comparator): Participants in the Active Comparator group will undergo a conventional strength training program using standard gym machines. Training sessions will occur 3 times per week for 12 weeks. The goal is to compare the outcomes of BioStrength training with traditional strength training.
  Interventions: Device: Conventional training
- BioStrength training (Experimental): Participants in the Intervention Group will undergo BioStrength training using Technogym equipment. The intervention will last for 12 weeks, with sessions conducted 3 times per week
  Interventions: Device: BioStrength Intervention

INTERVENTIONS:
Device: BioStrength Intervention — Participants in the Intervention Group will undergo BioStrength training using Technogym equipment. The intervention will last for 12 weeks, with sessions conducted 3 times per week
  Arms: BioStrength training
Device: Conventional training — Participants in the Active Comparator group will undergo a conventional strength training program using standard gym machines. Training sessions will occur 3 times per week for 12 weeks. The goal is to compare the outcomes of BioStrength training with traditional strength training.
  Arms: Control Group (No BioStrength Training)

SUMMARY:
This study aims to evaluate the effectiveness of Technogyms BioStrength equipment compared to traditional strength training equipment over a 12-week intervention period. The study will determine whether BioStrength machines produce more effective results in terms of muscle strength and body composition. Participants will be allocated to either the BioStrength group or the traditional training group using a minimisation technique to balance important prognostic factors such as handgrip strength, age and gender between the groups. Key measurements include maximum strength tests (10RM) for leg press and chest press, handgrip strength using a dynamometer, and body composition using bioimpedance analysis. Circumference measurements will also be taken. The study will assess whether BioStrength equipment provides superior results in muscle strength, body composition and training efficiency compared to conventional gym equipment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of Technogyms BioStrength machines compared to conventional strength training equipment in improving physical performance, muscle strength and body composition in untrained adults. The primary objective is to determine whether the BioStrength machines, which provide real-time feedback on movement amplitude, speed and force, lead to superior results in terms of muscle strength, body composition and training efficiency compared to conventional fitness equipment.

The study will follow a randomised controlled trial design over a 12-week period, using a minimisation technique to assign participants to either the BioStrength training group or the traditional strength training group. This technique ensures that key prognostic factors such as age, gender and baseline handgrip strength are balanced between the groups, as randomisation alone may not adequately address these factors in smaller sample sizes. Participants will attend three training sessions per week, each lasting approximately 60 minutes. The BioStrength group will use advanced machines that provide personalised feedback to optimise training, while the traditional group will use standard strength training machines without feedback technology.

The primary outcomes measured in this study include maximum strength, handgrip strength and body composition. Maximal strength will be assessed using the 10-RM (Repetition Maximum) test on leg press and chest press exercises, which determines the maximum weight participants can lift for 10 consecutive repetitions. Hand grip strength is measured using a Jamar dynamometer, with participants performing three attempts on each hand and recording the highest value. Body composition will be measured using bioimpedance analysis (BIA), a non-invasive method of estimating muscle mass and body fat percentage. In addition, circumference measurements of the arms, legs and waist will provide complementary data on changes in muscle growth and fat distribution.

The study will recruit 42 healthy adults aged 30-65 years with no more than six months of previous resistance training experience. Participants with a history of coronary heart disease, stroke, arthritis, or other medical conditions that could affect physical performance will be excluded. To allow for a 20% drop-out rate, the study will aim to recruit 21 participants per group. Recruitment will take place through a local fitness centre, using social media advertisements and flyers. Participants will be instructed to maintain their usual dietary habits throughout the 12-week intervention period. They will be asked not to make any significant changes to their diet or to introduce any new dietary supplements, as these could influence the outcomes related to muscle strength, body composition and overall physical fitness.

The study will consist of three phases: baseline, intervention and post-intervention. During baseline testing, participants will undergo strength and body composition assessments over two days, including the 10-RM test, handgrip strength measurements, BIA and circumference measurements. The intervention period will last 12 weeks, during which time participants will complete their assigned training programme under the supervision of a sports scientist who will conduct the assessments. After the intervention, all participants will repeat the same tests to assess changes in strength and body composition.

Data will be analysed using two-factor ANOVA to compare pre- and post-intervention outcomes between the two groups. The primary focus will be on changes in maximum strength, handgrip strength and body composition.

It is hypothesised that the BioStrength training group will show greater improvements in strength, handgrip strength and body composition compared to the traditional strength training group. The advanced feedback provided by the BioStrength machines is expected to result in more efficient and effective strength gains. This study has the potential to provide valuable insight into the benefits of using advanced strength training equipment and could influence future training protocols, particularly for individuals new to strength training.

The study has been approved by the Ethics Committee of the University of Graz and participants will be fully informed of the purpose, procedures and potential risks of the study before providing written informed consent. All data will be anonymised and confidentiality will be strictly maintained throughout the study.

This research could have significant implications for commercial fitness facilities as it aims to show whether BioStrength machines offer measurable benefits over traditional gym equipment. If successful, the study could contribute to the development of more efficient, data-driven training interventions that optimise muscle growth and body composition improvements for a wider population.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 30 and 65 years

  * Healthy individuals without significant medical conditions
  * Less than 6 months of prior strength training experience
  * Willing and able to participate in a 12-week training program
  * Capable of performing strength training exercises such as leg press and chest press
  * Able to provide written informed consent

Exclusion Criteria:

* • History of coronary heart disease

  * History of stroke
  * Need for changes in antihypertensive treatment within 3 months prior to study start
  * Arthritis
  * Pregnancy or less than three months postpartum
  * Pain and movement restrictions
  * Use of medications that affect muscle strength or performance (e.g., anabolic steroids, beta-2 agonists, glucocorticoids, statins, benzodiazepines, ACE inhibitors, angiotensin-II receptor blockers, diuretics)
  * Any medical condition preventing participation in planned endurance and strength training

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Mass | Baseline and Week 12
  Skeletal muscle mass will be measured using bioimpedance analysis (BIA) at baseline and after the 12-week intervention to evaluate changes in muscle mass.
Change in Body Fat Percentage | Baseline and Week 12
  Body fat percentage will be measured using bioimpedance analysis (BIA) at baseline and after the 12-week intervention to assess reductions in body fat.
Change in Handgrip Strength | Baseline and Week 12
  Handgrip strength will be measured using a Jamar dynamometer, with measurements taken at baseline and after the 12-week intervention.
Change in Maximal Strength (10-RM Test) | Baseline and Week 12
  Maximal strength will be measured using the 10-RM (Repetition Maximum) test for the leg press and chest press exercises at baseline and after the 12-week intervention.

SECONDARY OUTCOMES:
Customer Satisfaction (CSAT Questionnaire) | Week 2 and Week 12
  Customer satisfaction with the training experience will be measured using a standardized CSAT questionnaire at the end of the 12-week intervention.
Change in Circumference Measurements (Arm, Leg, and Waist) | Baseline and Week 12
  Circumference measurements of the arms, legs, and waist will be taken at baseline and after the 12-week intervention to assess changes in muscle size and fat distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Atia, Principal Investigator — University of Graz
Locations (1):
- CF Leibnitz, Leibnitz, Styria, Styria, Austria

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) used in the published results will be shared in an anonymized format. Access will be provided upon request through a secure data repository for researchers who meet the criteria for access to confidential data
Supporting Information: Study Protocol
Time Frame: Available upon publication for one year